CLINICAL TRIAL: NCT01180608
Title: Functional Imaging of the Therapeutic Effect of Pregabalin in Treatment for Neuropathic Pain in Patients With Diabetic Polyneuropathy Using Proton MR Spectroscopy
Brief Title: Functional Imaging of the Therapeutic Effect of Pregabalin in Treatment for Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Moens Maarten (Unknown)
Responsible Party: Maarten Moens, MD, UZ Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: vubmtmoensLIIRA
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Diabetic Neuropathies; Pain
Keywords: neuropathic pain; Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Neuralgia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Active Comparator)
  Interventions: Other: MR Spectroscopy
- placebo + pregabalin (Placebo Comparator)
  Interventions: Other: MR Spectroscopy

INTERVENTIONS:
Other: MR Spectroscopy — During each MR Spectroscopy session, we will measure at regions of interest (rACC, both thalami, dominant DLPC) the levels of the following biochemical substances:
  * gamma-aminobutyric acid (GABA)
  * glutamate (Glu)
  * glutamine (Gln)
  * N-acetylaspartate (NAA)
  * Choline-containing compounds (Cho)
  * Creatine plus phophocreatine (total creatine: Cr)
  * Myo-inositiol (Ins)
  * Choline (Cho)
  * Glucose (Glc)
  * Lactate (Lac)

SUMMARY:
Functional Imaging of the therapeutic effect of Pregabalin in treatment for neuropathic pain in patients with Diabetic Polyneuropathy using proton Magnetic Resonance Spectroscopy (MRS):

The aim of our study is to investigate the effect of Pregabalin as a treatment for neuropathic pain in a homogeneous study population, using proton MRS (1H MRS) focusing on four regions of interest (bilateral thalami, rostral anterior cingulated cortex (rACC) and dominant dorsolateral prefrontal cortex (DLPC).

DETAILED DESCRIPTION:
spectrum measurements at: thalamus left thalamus right rostral anterior cingulated cortex dominant dorsolateral prefrontal cortex

measurements: gamma-aminobutyric acid (GABA) glutamate (Glu) glutamine (Gln) N-acetylaspartate (NAA) Choline-containing compounds (Cho) Creatine plus phophocreatine (total creatine: Cr) Myo-inositiol (Ins) Choline (Cho) Glucose (Glc) Lactate (Lac)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with painful DPN
* Patient willing to provide informed consent
* Type 1 or type 2 diabetes with HbA1c ≤ 11%
* Stable antidiabetic medication for 30 days prior to randomization
* Duration of painful DPN ≥ 3 months
* Visual analogue scale (VAS) score ≥ 4

Exclusion Criteria:

* Creatinine clearance ≤ 60mL/min
* Presence of other clinically significant or disabling chronic pain condition
* Active malignancy
* Evidence of an active disruptive psychiatric disorder or other known condition that might influence the perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by the investigator
* Life expectancy less than 1 year
* Existing or planned pregnancy
* Extreme fear for entering MRI
* General contraindication for MRI (pacemaker, etc…)
* Patients participating in other clinical trials
* Age <18 years
* Prior use of potential retinotoxins
* Prohibited medications without proper wash-out period (>7days, depending on the type of medication):

  * medications and supplements commonly used for relief of neuropathic pain
  * antiepileptics
  * antidepressants (except for stable regiments of SSRIs for treatment of anxiety or depression)
  * NSAID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
cerebral neurobiological effect of pregabaline as treatment for neuropathic pain | 1 year
  We will measure changes in neurotransmitter levels in the brain (gamma-aminobutyric acid (GABA) glutamate (Glu) glutamine (Gln) N-acetylaspartate (NAA) Choline-containing compounds (Cho) Creatine plus phophocreatine (total creatine: Cr) Myo-inositiol (Ins) Choline (Cho) Glucose (Glc) Lactate (Lac)) before and after treatment with pregabaline. Specific interest in ratio GABA/Gln and GABA/Glu: relationship between inhibitory and excitatory neurotransmittors

SECONDARY OUTCOMES:
cerebral neurobiological changes in relationship with dose dependent therapeutic effect of treatment with pregabaline | 1 year
  A possible dose dependent effect of treatment with Pregabalin on cerebral neurochemical changes (gamma-aminobutyric acid (GABA) glutamate (Glu) glutamine (Gln) N-acetylaspartate (NAA) Choline-containing compounds (Cho) Creatine plus phophocreatine (total creatine: Cr) Myo-inositiol (Ins) Choline (Cho) Glucose (Glc) Lactate (Lac)) and clinical effects (pain and quality of life scales) will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Derived] De Jaeger M, Goudman L, Van Schuerbeek P, De Mey J, Keymeulen B, Brouns R, Moens M. Cerebral Biochemical Effect of Pregabalin in Patients with Painful Diabetic Neuropathy: A Randomized Controlled Trial. Diabetes Ther. 2018 Aug;9(4):1591-1604. doi: 10.1007/s13300-018-0460-y. Epub 2018 Jun 27. PMID 29951977